CLINICAL TRIAL: NCT02352818
Title: Chronic Total Occlusion Registry
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57285
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Total Coronary Occlusions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no study intervention

SUMMARY:
The aim of this CTO registry is to gather data including patient demographic date, cardiac risk factors, procedural technical data and procedural success/outcome rates. Furthermore, we aim to evaluate the safety and performance of various CTO specific guidewires, devices (such as the CrossBoss/Stingray dissection re-entry device) and other recognised and approved techniques (retrograde wire escalation, retrograde dissection re-entry techniques). The incidence of recognized complications (dissections, perforations, cardiac tamponade, vascular complications, radiation injury, acute kidney injury) will also evaluated. The investigator will assess clinical outcome at 1 year after successful CTO procedures.

DETAILED DESCRIPTION:
This objectives of this single-center CTO registry are to:

1. Gather prospective clinical data on all consecutive patients undergoing complex difficult CTO PCI procedures including patient demographic date, cardiac risk factors, procedural technical data (contrast volume, radiation exposure, procedure time and procedural success/outcome rates.
2. Evaluate the safety and performance of various CTO dedicated guidewires, devices (such as the CrossBoss/Stingray anterior dissection re-entry device) and other recognised and approved techniques (retrograde wire escalation, retrograde dissection re-entry techniques).
3. Evaluate the incidence and severity of recognized complications such as coronary dissections, coronary perforations (+/- need for emergency pericardiocentesis), acute kidney injury, radiation injury, access site vascular complications.
4. Evaluate the medium-term outcome (recurrence of symptoms, major cardiovascular events (cardiac death, myocardial infarction, target lesion revascularization, target vessel revascularization) during a routine out-patient consultation (planned as part of normal standard care) at 1 year post successful CTO PCI. After this consultation, the patient may choose to have cardiology follow-up at the UZ Leuven or with his/her referring cardiologist.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing an elective attempt at percutaneous revascularization of a chronic total occlusion are eligible for inclusion in the CTO registry. A chronic total occlusion is defined as an occluded coronary artery with TIMI 0 flow that has been occluded for 3 months or more. By definition all patients will have been judged to be acceptable candidates for an attempt at revascularization before consenting to be part of the CTO registry.

Exclusion Criteria:

* There are no specific exclusion criteria. If the patient does not wish to consent to having his personal data kept in a registry the patient will not be included in the CTO registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing percutaneous attempt at revascularisation of a chronic total coronary occlusion
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-01-26; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Succes rate of procedure | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiovascular Disease, University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided